CLINICAL TRIAL: NCT01427881
Title: A Phase II Study to Evaluate the Efficacy of Posttransplant Cyclophosphamide for Prevention of Chronic Graft-versus-Host Disease After Allogeneic Peripheral Blood Stem Cell Transplantation
Brief Title: Cyclophosphamide for Prevention of Graft-Versus-Host Disease After Allogeneic Peripheral Blood Stem Cell Transplantation in Patients With Hematological Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marco Mielcarek, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2541.00; NCI-2011-02459 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH)
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Myeloid Leukemia in Remission; Adult Erythroleukemia (M6a); Adult Nasal Type Extranodal NK/T-cell Lymphoma; Adult Pure Erythroid Leukemia (M6b); Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Blastic Phase Chronic Myelogenous Leukemia; Childhood Acute Erythroleukemia (M6); Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Megakaryocytic Leukemia (M7); Childhood Acute Myeloid Leukemia in Remission; Childhood Burkitt Lymphoma; Childhood Chronic Myelogenous Leukemia; Childhood Diffuse Large Cell Lymphoma; Childhood Immunoblastic Large Cell Lymphoma; Childhood Myelodysplastic Syndromes; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Chronic Myelomonocytic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; Cutaneous B-cell Non-Hodgkin Lymphoma; de Novo Myelodysplastic Syndromes; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Philadelphia Chromosome Negative Chronic Myelogenous Leukemia; Post-transplant Lymphoproliferative Disorder; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage III Multiple Myeloma; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Megakaryoblastic, Acute; Leukemia, Erythroblastic, Acute; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Blast Crisis; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Cyclophosphamide; Cyclosporine; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation; fludarabine phosphate; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (TBI, PBSCT, and cyclophosphamide GVHD prophylaxis) (Experimental): PREPARATIVE REGIMEN: Patients receive TBI BID on days -4 or -3 to -1. Some patients also receive fludarabine IV daily on days -5 to -2 and busulfan IV over 3 hours QD or over 2 hours every 6 hours on days -5 to -2. Patients may also undergo CNS prophylaxis, testicular irradiation, and/or involved field irradiation as per standard practice.
  TRANSPLANTATION: Patients undergo allogeneic PBSCT on day 0 per standard practice.
  GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 1-2 hours on days 3-4. Patients also receive cyclosporine IV every 12 hours or every 8 hours beginning on day 5 with taper on days 56-126.
  Interventions: Drug: cyclophosphamide; Drug: cyclosporine; Procedure: peripheral blood stem cell transplantation; Radiation: total-body irradiation; Drug: fludarabine phosphate; Drug: busulfan; Procedure: allogeneic hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: cyclosporine — Given IV
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Procedure: peripheral blood stem cell transplantation — Undergo allogeneic PBSCT
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: busulfan — Given IV
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic PBSCT

SUMMARY:
This phase II trial studies how well cyclophosphamide works in preventing chronic graft-versus-host disease after allogeneic peripheral blood stem cell transplant in patients with hematological malignancies. Giving chemotherapy and total-body irradiation before transplantation helps stop the growth of cancer cells and prevents the patient's immune system from rejecting the donor's stem cells. Healthy stem cells from a donor that are infused into the patient help the patient's bone marrow make blood cells; red blood cells, white blood cells, and platelets. Sometimes, however, the transplanted donor cells can cause an immune response against the body's normal cells, which is called graft-versus-host disease (GVHD). Giving cyclophosphamide after transplant may prevent this from happening or may make chronic GVHD less severe.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary objective of this study is to assess outcomes when high-dose cyclophosphamide (CY) is administered on days 3 and 4 followed by cyclosporine (CSP) after human leukocyte antigen (HLA)-matched related or unrelated mobilized blood cell transplantation with total-body irradiation (TBI) or busulfan (BU)-based conditioning.

SECONDARY OBJECTIVES:

I. The secondary objective of this study is to assess hematopoietic cell transplantation (HCT) outcomes when withdrawal of CSP is accelerated in patients without acute graft-versus-host disease (GVHD).

OUTLINE: Patients' conditioning regimens are determined by the Clinical Coordinator after consultation with the attending physician. Based on disease, patients receive either TBI or fludarabine and busulfan.

PREPARATIVE REGIMEN: Patients receive TBI twice daily (BID) on days -4 or -3 to -1. Some patients also receive fludarabine intravenously (IV) daily on days -5 to -2 and busulfan IV over 3 hours once daily (QD) or over 2 hours every 6 hours on days -5 to -2. Patients may also undergo central nervous system (CNS) prophylaxis, testicular irradiation, and/or involved field irradiation as per standard practice.

TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplantation (PBSCT) on day 0 per standard practice.

GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 1-2 hours on days 3-4. Patients also receive cyclosporine IV every 12 hours or every 8 hours beginning on day 5 with taper on days 56-126.

Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at day 180 and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphocytic leukemia (ALL) in morphologic first complete remission (CR1) with high risk features defined as, but not limited to: evidence of adverse cytogenetics such as t(9;22), t(1;19), t(4;11), or mixed-lineage leukemia (MLL) rearrangements; presence of minimal residual disease; progenitor B-cell immunophenotype; high white blood cells (WBC) at diagnosis (> 30,000/ul in B-ALL; > 100,000/ul in T-ALL); or delayed attainment of CR (> 4 weeks) after induction therapy; additional clinical characteristics deemed to confer a high relapse risk may be discussed with and approved by the Principal Investigator (PI)
* Acute myeloid leukemia (AML) in CR1 EXCEPT patients with low-risk features defined as:

  * Inv 16 or t(8;21) in the absence of c-kit mutations
  * Normal karyotype who are FLT3-ITD-negative and NPM1-positive in the absence of c-kit mutations
  * Patients with respective "low-risk" features are eligible, however, if (i) more than 1 cycle of induction therapy was required to achieve CR1 (ii) the patient had a preceding myelodysplastic syndrome (MDS) other than myelofibrosis, or (iii) secondary AML
* Acute leukemia in 2nd or greater CR (CR >= 2)
* Refractory or relapsed AML with =< 10% bone marrow blasts and no circulating blasts or proven extramedullary disease
* AML transformed from myelodysplastic syndrome (MDS) with < 10% bone marrow blasts
* MDS with following high risk features:

  * High risk cytogenetics (including, but not limited to: 7q--, inv[3], t[3q], del[3q] or complex karyotype)
  * International Prognostic Scoring System (IPSS) intermediate (INT)-2 or greater
  * Treatment-related MDS
  * Any phase of MDS if patient is < 21 years of age
* Chronic myelogenous leukemia (CML) beyond 1st chronic phase or resistant or intolerant to tyrosine kinase inhibitors (adults) or any phase (pediatric < 21 years)
* Chronic myelomonocytic leukemia
* Philadelphia-negative myeloproliferative disorder
* Lymphoma: relapsed chemotherapy-sensitive (complete or partial response) Hodgkin or non-Hodgkin lymphoma
* Multiple myeloma-stage III
* The patient or legal representative must be able to understand and give written informed consent
* DONORS: The donor must be a genotypically HLA-identical sibling, a phenotypically HLA-matched first-degree relative, or an unrelated donor who is molecularly matched with the patient at HLA-A, B, C, DRB1
* DONORS: Donors must meet the selection criteria for administration of G-CSF (filgrastim) and apheresis defined by the Foundation for the Accreditation of Cell Therapy (FACT) and will be screened per the American Association of Blood Banks (AABB)
* DONORS: Donors must be capable of giving informed consent

Exclusion Criteria:

* Prior autologous or allogeneic stem cell transplant
* Performance status > 2 (Eastern Cooperative Oncology Group [ECOG]) or < 50 (Lansky; for patients < 16 years old)
* Uncontrolled infection; the protocol principal investigator (PI) will be final arbiter if there is uncertainty regarding whether a previous infection is under adequate control to allow enrollment in the study
* Positive serology for human immunodeficiency virus (HIV)-1, 2 or human T cell lymphotropic virus (HTLV)-1, 2
* Left ventricular ejection fraction < 45% or shortening fraction < 25%; no uncontrolled arrhythmias or symptomatic cardiac disease
* Symptomatic pulmonary disease; forced expiratory volume in one second (FEV1), forced vital capacity (FVC), diffusion capacity of the lung for carbon monoxide (DLCO) =< 50% of predicted (corrected for hemoglobin); if pulmonary function tests cannot be performed, an oxygen saturation < 92% on room air
* Calculated (Cockcroft-Gault or appropriate calculation for pediatric patients) serum creatinine clearance =< 60 mL/min; if the calculated CrCl is 50-60 mL/min, but a measured CrCl by 24 hour urine collection is > 60 mL/min, this measurement is acceptable
* Total serum bilirubin more than twice upper normal limit
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) more than 3-fold higher than laboratory upper normal limits
* Female patient must have negative serum pregnancy test (all women of child bearing-potential must have test performed)
* DONORS: Potential donors who for psychological, physiological, or medical reasons cannot tolerate administration of G-CSF or apheresis
* DONORS: Donors who are allergic to filgrastim or Escherichia (E.) coli-derived proteins
* DONORS: Donor-related risks to recipients
* DONORS: Positive anti-donor lymphocytotoxic crossmatch
* DONORS: Donors who are positive for HIV

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-09; Primary Completion 2014-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Mielcarek, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Mielcarek M, Furlong T, O'Donnell PV, Storer BE, McCune JS, Storb R, Carpenter PA, Flowers ME, Appelbaum FR, Martin PJ. Posttransplantation cyclophosphamide for prevention of graft-versus-host disease after HLA-matched mobilized blood cell transplantation. Blood. 2016 Mar 17;127(11):1502-8. doi: 10.1182/blood-2015-10-672071. Epub 2016 Jan 13. PMID 26764356

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (TBI, PBSCT, and Cyclophosphamide GVHD Prophylaxis): PREPARATIVE REGIMEN: Patients receive TBI BID on days -4 or -3 to -1. Some patients also receive fludarabine IV daily on days -5 to -2 and busulfan IV over 3 hours QD or over 2 hours every 6 hours on days -5 to -2. Patients may also undergo CNS prophylaxis, testicular irradiation, and/or involved field irradiation as per standard practice.
  TRANSPLANTATION: Patients undergo allogeneic PBSCT on day 0 per standard practice.
  GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 1-2 hours on days 3-4. Patients also receive cyclosporine IV every 12 hours or every 8 hours beginning on day 5 with taper on days 56-126.
  cyclophosphamide: Given IV
  cyclosporine: Given IV
  peripheral blood stem cell transplantation: Undergo allogeneic PBSCT
  total-body irradiation: Undergo TBI
  fludarabine phosphate: Given IV
  busulfan: Given IV
  allogeneic hematopoietic stem cell transplantation: Undergo allogeneic PBSCT
Period: Overall Study
Arm/Group | Treatment (TBI, PBSCT, and Cyclophosphamide GVHD Prophylaxis)
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (TBI, PBSCT, and Cyclophosphamide GVHD Prophylaxis)
Number analyzed (Participants) | 43
Age, Continuous [Median (Full Range); unit: years] | 38 [3 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Chronic GVHD Requiring Systemic Immunosuppressive Treatment
Description: Chronic GVHD will be defined by National Institutes of Health (NIH) criteria and requiring systemic treatment. A reduction in the cumulative incidence of GVHD from ~35% to ~15% at 1 year would represent a reasonable goal. A sample size of 42 patients provides 90% power to observe such a difference with one-side 5% type-1 error.
Time Frame: At 1 year after transplantation
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Treatment (TBI, PBSCT, and Cyclophosphamide GVHD Prophylaxis)
Number analyzed (Participants) | 43
percent of patients | 16 [5 to 28]

2. Secondary Outcome: Donor Engraftment
Description: Donor engraftment is defined as the count (percent) of patients with full donor chimerism. Full donor chimerism is defined as at least 95% donor CD3 cells in peripheral blood.
Time Frame: At day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (TBI, PBSCT, and Cyclophosphamide GVHD Prophylaxis)
Number analyzed (Participants) | 43
Participants | 6

3. Secondary Outcome: Grades II-IV and III-IV Acute GVHD
Description: Grades II-IV and III-IV GVHD will be assessed with the use of cumulative incidence plots.
Time Frame: Through day +100 post-transplant
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (TBI, PBSCT, and Cyclophosphamide GVHD Prophylaxis)
Number analyzed (Participants) | 43
percentage of patients
  Grades II-IV GVHD | 77
  Grades III-IV GVHD | 0

4. Secondary Outcome: Duration of Systemic Immunosuppressive Treatment
Description: The need for additional immunosuppressive treatment with agents other than those used for prophylaxis, the reasons for their administration (acute GVHD, chronic GVHD, or other reasons) and the duration of its administration will be determined. Patients will be monitored to determine the duration of systemic immunosuppressive treatment. Primary and secondary treatment of acute GVHD and withdrawal of systemic immunosuppressive treatment will be assessed with the use of cumulative incidence plots.
Time Frame: Up to 5 years
Population: This data was not collected.
Arm/Group | Treatment (TBI, PBSCT, and Cyclophosphamide GVHD Prophylaxis)
Number analyzed (Participants) | 0

5. Secondary Outcome: Persistent or Recurrent Malignancy After HCT
Description: Recurrent or progressive malignancy will be assessed with the use of cumulative incidence plots. Recurrent malignancy will be defined by hematologic criteria. Recurrent malignancy will also be defined as any unplanned medical intervention designed to prevent progression of malignant disease in patients who have molecular, cytogenetic or flow-cytometric evidence of malignant cells after transplantation.
Time Frame: At 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (TBI, PBSCT, and Cyclophosphamide GVHD Prophylaxis)
Number analyzed (Participants) | 43
percentage of patients | 17 [5 to 29]

6. Secondary Outcome: Non-relapse Mortality
Description: Defined as death in the absence of recurrent or progressive malignancy after HCT. Non-relapse morality will be assessed with the use of cumulative incidence plots. This secondary endpoint will be characterized and presented as a cumulative incidence.
Time Frame: At 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (TBI, PBSCT, and Cyclophosphamide GVHD Prophylaxis)
Number analyzed (Participants) | 43
percentage of patients | 14 [4 to 25]

7. Secondary Outcome: Overall Survival
Description: Overall survival will be evaluated as Kaplan-Meier estimates.
Time Frame: At 1 year post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (TBI, PBSCT, and Cyclophosphamide GVHD Prophylaxis)
Number analyzed (Participants) | 43
percentage of patients | 75.6 [63.5 to 90.1]

8. Secondary Outcome: Disease-free Survival
Description: Disease-free survival will be evaluated as Kaplan-Meier estimates.
Time Frame: At 1 year post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (TBI, PBSCT, and Cyclophosphamide GVHD Prophylaxis)
Number analyzed (Participants) | 43
percentage of patients | 73.8 [61.6 to 88.5]

9. Secondary Outcome: Hematologic Recovery
Description: Descriptive statistics will be used to assess the median days of neutrophil and platelet recovery. The day of neutrophil recovery is defined as the first day of three consecutive lab values on different days, after the conditioning regimen-induced nadir of blood counts, that the absolute neutrophil count is > 500/uL. The day of platelet recovery is defined as the first day of three consecutive lab values on different days, after the conditioning regimen-induced nadir of blood counts, that the platelet count is >= 20,000/uL without platelet transfusion support in the seven days prior.
Time Frame: Up to day +100
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (TBI, PBSCT, and Cyclophosphamide GVHD Prophylaxis)
Number analyzed (Participants) | 43
days
  Neutrophil Engraftment | 19 [16 to 37]
  Platelet Engraftment | 14 [10 to 47]

10. Secondary Outcome: Graft Failure
Description: Descriptive statistics will be used to assess the incidence of primary graft failure and secondary graft failure. Primary graft failure is defined as failure to achieve a sustained neutrophil count of >= 500/uL by >= 28 days post-transplant. Secondary graft failure is defined as the decline in neutrophil count to < 500/uL after achieving engraftment which is unrelated to infection or drug effect and is unresponsive to stimulation by growth factors.
Time Frame: By greater than or equal to 28 days post-transplant
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (TBI, PBSCT, and Cyclophosphamide GVHD Prophylaxis)
Number analyzed (Participants) | 43
percentage of patients | 2

ADVERSE EVENTS:
Time Frame: For all-cause mortality: 1 year after transplant For adverse events and serious adverse events, not mortality, will be monitored and recorded through the time of discharge from the transplant center
Arm/Group | Treatment (TBI, PBSCT, and Cyclophosphamide GVHD Prophylaxis)
All-Cause Mortality (participants affected / at risk) | 11/43
Serious Adverse Events (participants affected / at risk) | 22/43
Other Adverse Events (participants affected / at risk) | 40/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment (TBI, PBSCT, and Cyclophosphamide GVHD Prophylaxis) (N=43)
Infection/Fever (Blood and lymphatic system disorders) | 13 (18) — Various organs (blood, pulmonary, bladder, etc)
Disease recurrence/MRD (Blood and lymphatic system disorders) | 4 (4)
Bradycardia (Cardiac disorders) | 1 (1)
Delayed engraftment (Blood and lymphatic system disorders) | 1 (1)
Graft failure/poor graft function (Blood and lymphatic system disorders) | 1/1 (2)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
GVHD (Immune system disorders) | 6 (7)
Respiratory (not infection) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
RS3PE (rheumatologic) (Musculoskeletal and connective tissue disorders) | 1 (1)
Orthastic hypotension (Vascular disorders) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (TBI, PBSCT, and Cyclophosphamide GVHD Prophylaxis) (N=43)
Failure to engraft by day 28 (Blood and lymphatic system disorders) | 3 (3)
Persistent n/v thru day 28 and not related to GVHD (Gastrointestinal disorders) | 3 (3)
Heart failure or LV dysfunction (grade 3-5) (Cardiac disorders) | 0 (0)
Mucositis (grade 3-5; requiring TPN) (Gastrointestinal disorders) | 40 (40)
Cystitis or hematuria (grade 2-5; not infection) (Renal and urinary disorders) | 1 (1)
Other (grade 3-5) (General disorders) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes